CLINICAL TRIAL: NCT00125671
Title: A Phase III Randomized Trial of Warfarin Plus Antiplatelet Therapy Versus Antiplatelet Therapy Alone in Patients With Peripheral Vascular Disease
Brief Title: Warfarin and Antiplatelet Vascular Evaluation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anand, Sonia, M.D. (Individual)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Ontario (Other)
Organization: Warfarin and Antiplatelet Vascular Evaluation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCT-37413; T4913
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-09

CONDITIONS: Peripheral Vascular Diseases; Cardiovascular Diseases
Keywords: Warfarin and Antiplatelet Vascular Evaluation; Peripheral vascular disease; Atherosclerosis; cardiovascular events; Ischemia; oral anticoagulants; low ankle-brachial index; moderate intensity warfarin; International normalized ratio [INR]
MeSH Terms: conditions — Peripheral Vascular Diseases; Cardiovascular Diseases; Atherosclerosis; Ischemia | interventions — Warfarin

INTERVENTIONS:
Drug: Warfarin

SUMMARY:
The purpose of this study is to evaluate whether the addition of warfarin (a blood-thinning medication) to an antiplatelet therapy like aspirin is better than antiplatelet therapy alone (i.e. usual treatment) for the prevention of leg surgery, heart attacks, stroke and death in people with peripheral vascular disease.

DETAILED DESCRIPTION:
Atherosclerosis is the underlying cause of peripheral vascular disease (PVD) of the lower extremities, and leads to intermittent claudication, leg ulceration and gangrene. More importantly, symptomatic PVD is an ominous sign that widespread atherosclerosis is present and patients with this condition suffer a threefold increase in myocardial infarction (MI), stroke, and CV death. These CV events are a consequence of rupture of an atherosclerotic plaque, which leads to platelet activation and thrombin generation, thrombus formation and occlusion of a critical blood vessel. Antiplatelet therapy has been clearly demonstrated to reduce major CV events. It is also reasonable to expect that this process may be further attenuated by the addition of an anti-thrombin agent (such as warfarin) in combination with antiplatelet agents.

WAVE is a large, international, multicentre, randomized clinical trial in high-risk PVD patients to evaluate the additional benefit of moderate intensity warfarin (target INR of 2.4-3.0) to antiplatelet therapy compared to antiplatelet therapy alone in reducing serious cardiovascular events.

There are currently 80 active centres following participants in Canada, Poland, Australia, Hungary, China, Ukraine, and the Netherlands. Following randomization to one of the two treatment groups, participants will require clinic or phone follow-up visits every 3 months for 2.5 or 3.5 years. For participants on warfarin, INRs will be measured monthly or more frequently if required. For participants who stop warfarin therapy prematurely, every attempt will be made to have them restart it

ELIGIBILITY:
Inclusion Criteria:

* Intermittent claudication with objective evidence of PVD (e.g. ankle-brachial index [ABI] < 0.90)
* Ischemic rest pain of the lower limbs
* Ischemic non-healing ulcers or focal gangrene
* Amputation for vascular causes
* Previous peripheral vascular revascularization (angioplasty or bypass surgery)
* Blue toe syndrome
* Other significant peripheral arterial disease (e.g. carotid stenosis)
* Vascular disease and evidence of asymptomatic peripheral arterial disease [PAD] (i.e. ABI < 0.90)

Exclusion Criteria:

Temporary:

* Potential subjects will be temporarily excluded if they need to undergo:

  * vascular diagnostic (angiography) or interventional procedures (arterial bypass graft surgery or angioplasty); or
  * limb amputation for vascular insufficiency.

Permanent:

* Subjects will be excluded for the following:

  * active bleeding or high risk bleeding;
  * clear indication for long-term warfarin use (i.e. atrial fibrillation);
  * previous allergy or intolerance to warfarin;
  * stroke in the last 6 months;
  * renal failure requiring dialysis;
  * known significant abdominal aortic or cerebral aneurysm;
  * peripheral arterial aneurysms (iliac or femoral) without evidence of lower limb ischemia;
  * significant liver disease (i.e. cirrhosis);
  * cancer with a life expectancy < 6 months;
  * anticipated non-adherence to warfarin;
  * excessive alcohol use;
  * pregnancy or planning to become pregnant; or
  * failure to provide informed consent.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400
Dates: Start 2000-01; Study Completion 2006-04

PRIMARY OUTCOMES:
The composite of cardiovascular (CV) death, first occurrence of myocardial infarction (MI), or stroke
The composite of CV death, first occurrence of MI, stroke, or severe ischemia requiring urgent intervention of the coronary (PTCA, CABG) or peripheral artery circulation (thrombolytic therapy, angioplasty, bypass surgery, limb amputation)

SECONDARY OUTCOMES:
CV death, MI, stroke, amputation, revascularization of the coronary or peripheral arteries, or admission to hospital for unstable angina with electrocardiogram (ECG) changes
CV death, MI, stroke, transient ischemic attack (TIA), amputation or revascularization of the coronary, carotid, or leg arteries
All cause death, MI, TIA, stroke, amputation, or revascularization of the coronary or peripheral arteries

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Anand, MD PhD FRCPc, Principal Investigator — Population Health Research Institute, McMaster University
Locations (1):
- Population Health Research Institute, McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Background] WAVE Investigators. The effects of oral anticoagulants in patients with peripheral arterial disease: rationale, design, and baseline characteristics of the Warfarin and Antiplatelet Vascular Evaluation (WAVE) trial, including a meta-analysis of trials. Am Heart J. 2006 Jan;151(1):1-9. doi: 10.1016/j.ahj.2005.03.021. PMID 16368284
- [Derived] Warfarin Antiplatelet Vascular Evaluation Trial Investigators; Anand S, Yusuf S, Xie C, Pogue J, Eikelboom J, Budaj A, Sussex B, Liu L, Guzman R, Cina C, Crowell R, Keltai M, Gosselin G. Oral anticoagulant and antiplatelet therapy and peripheral arterial disease. N Engl J Med. 2007 Jul 19;357(3):217-27. doi: 10.1056/NEJMoa065959. PMID 17634457